CLINICAL TRIAL: NCT05768802
Title: Evaluation of an Implantable Intramuscular Device to Control a Myoelectric Prosthesis
Brief Title: Evaluation of Myoelectric Implantable Recording Array (MIRA) in Participants With Transradial Amputation
Acronym: MIRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boninger, Michael, MD (Other)
Collaborators: Ripple Therapeutics Corporation (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Robert Gaunt, PhD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY21040146; 1U44NS123301-01 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-03-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Amputation; Amputation; Traumatic, Hand
Keywords: hand amputation; wrist amputation; transradial amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MIRA Device (Experimental): All participants enrolled in the study and who meet eligibility criteria will be implanted with the MIRA device in their residual limb. There is no control group.
  Interventions: Device: Myoelectric Implantable Recording Array (MIRA)

INTERVENTIONS:
Device: Myoelectric Implantable Recording Array (MIRA) — The Myoelectric Implantable Recording Array (MIRA) will use electromyography to detect the electrical activity of forearm muscles and transmit that information to an externally-powered prosthetic limb. The MIRA is implanted under the skin.

SUMMARY:
The purpose of this research study is to see how well a new type of myoelectric prosthesis works. A myoelectric prosthesis is a robotic limb for amputees that is controlled by sensing the activity of muscles in the body above the amputation level. This study involves a medical procedure to implant the Myoelectric Implantable Recording Array (MIRA) in the residual limb. The procedure will be performed under sedation by a physician. When muscles contract, they generate an electrical signal that can be sensed by MIRA and used to control the prosthetic limb. Myoelectric prosthetic limbs normally use electrodes that are placed on the surface of the skin to control different movements. However, MIRA is implanted under the skin, which could improve the ability to control the myoelectric prosthesis. After the MIRA is implanted, training will occur to learn how to control the prosthesis using the muscles in the residual limb. The device can stay implanted for up to one year. The device will be removed (explanted) by a physician.

DETAILED DESCRIPTION:
A well-documented challenge with current myoelectric devices is the common use of only two surface EMG electrodes to record control signals, typically one on each of the extensor and flexor muscle compartments in the residual limb. With this electrode configuration, just a single motion can be controlled at any given time. Changing to new motions or grasp patterns typically requires a secondary switching method. This sequential control enables pre-programmed functional grasps, and can be selected by patterns of co-contraction of antagonist muscle groups. However, this approach has limited success due to the slow and non-intuitive nature of the required muscular activations. For example, contraction of flexor muscles may be used to close the hand, but in order to rotate the wrist, a co-contraction of the flexors and extensors (to switch control modes) followed by flexor contraction is required. This non-intuitive approach ignores the normal function of forearm muscles and has a further disadvantage that simultaneous control of hand aperture and wrist rotation is impossible. Adding additional grasping patterns can make the problem worse and often requires the user to step through the different pre-programmed patterns by making multiple co-contractions until the correct movement is selected. Surface electrode-based systems also rely on strong muscle contractions, which are inefficient and contribute to awkward usability and ultimate rejection of the prosthesis. Other complications that are associated with surface electrodes are signal changes due to environmental conditions such as sweating, daily changing of electrode locations due to skin-related issues, and susceptibility to crosstalk and movement artifacts. In contrast, implantable electrodes are protected from environmental conditions, remain fixed in place, can record small signals from gently contracting muscles, and can record many different signals to potentially allow for more complex and simultaneous control of multiple joints.

Recent research with myoelectric control has focused on developing new control paradigms, such as simultaneous multi-degree of freedom control and proportional velocity control. Often, surface EMG recordings from an antagonistic pair of muscles are used to control a single degree of freedom. Implantable electrodes have shown promise as an alternative method in preliminary human subject studies, and recent research has demonstrated that up to three degrees-of-freedom have been simultaneously controlled in a virtual environment using intramuscular electrodes, as well as proportional velocity control. The Implantable Myoelectric Sensor (IMES®) System utilizes eight implanted electrodes (six actively needed for control, two as back-ups) to control three degrees-of-freedom. Another study using the same EMG leads and electrode configuration as MIRA, implanted percutaneously, enabled simultaneous control of up to 6 degrees of freedom (thumb flexion, index flexion, middle flexion, thumb adduction and abduction, wrist flexion and extension, and wrist pronation and supination) of an advanced prosthesis. As myoelectric prostheses move away from preprogrammed movements and pattern recognition, a minimum of two electrodes implanted in separate muscle targets appears to be necessary to control a single degree of freedom.

The investigator's approach aims to address the limitations of controlling state-of-the-art prosthetic hands. Multichannel intramuscular EMG recordings using the MIRA implant will be used to drive simultaneous hand and wrist movements providing a significant improvement in motor control over the current state-of-the-art. More specifically, the goal is to achieve control of wrist rotation and open/close of the hand and optimally, flexion/extension of the wrist and independent flexion/extension of four fingers. People with transradial amputations will be recruited into this study with the goal of restoring hand and wrist function.

The investigators have designed MIRA to eliminate percutaneous connections, which will reduce the risk of infection and minimize the amount of care required by study subjects. The study is designed to last for one year including a significant amount of in-home testing. Telerehabilitation principles (e.g. remote monitoring, regular progress checks) will be used to ensure frequent communication with investigators and regular assessment of device performance. Conducting a year-long study will provide sufficient time to allow for subjects to learn to use their new device and also allow us to document long-term device performance. The investigators will collect preliminary safety data and document the type and frequency of any adverse events that occur for the duration of the implantation. EMG signal quality and overall device performance over the duration of the implantation will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a unilateral transradial amputation or wrist disarticulation.
2. Subjects must demonstrate independent voluntary control of muscles in the flexor and extensor compartments of the forearm
3. Subjects must be over 1-year post-amputation at time of implantation.
4. Subjects must be between the ages of 22 and 70 years old. Subjects outside this age range may be at an increased surgical risk and increased risk of fatigue during prosthetic training.
5. Subjects must be able to communicate with the investigators in English because of the need to follow the instructions of the study team.
6. Subjects must show an understanding of the study goals and have the ability to follow simple directions as judged by the investigators.
7. Subjects must pass a neuropsychological and psychosocial assessment.
8. Documentation of informed consent must be obtained from the subject.

Exclusion Criteria:

1. Subjects must be able to function without the use of a prosthesis, or have access to assistance, for a period of 6 weeks following implantation and explantation surgeries.
2. Subjects must not have visual impairment such that extended viewing of a computer monitor would be difficult even with ordinary corrective lenses.
3. Subjects who have another serious disease(s) or disorder(s) that could affect their ability to participate in this study (verified during pre-op anesthesia evaluation to determine surgical risk status) will be excluded.
4. Subjects must not have phantom limb pain that is self-reported to be severe (options are no pain, mild pain, moderate pain, severe pain).
5. Subjects must not have any type of implantable generator such as a pacemaker, spinal cord stimulator, cochlear implant, deep brain stimulator (DBS) or DBS leads, vagus nerve stimulator, or defibrillator.
6. Female subjects of childbearing age must not be pregnant, lactating, or plan to become pregnant during the next 25 months.
7. Subjects must have no history of peripheral vascular disease that could impact wound healing.
8. Subjects who require routine MRI, therapeutic ultrasound, or diathermy as part of their ongoing care will be excluded.
9. Subjects must not have osteomyelitis.
10. Subjects must have no history of intractable clinically relevant cardiac arrhythmias.
11. Subjects must have no active infection(s) or unexplained fever(s) (verified during pre-op anesthesia evaluation to determine surgical risk status).
12. Subject must have no history of ongoing untreated alcoholism.
13. Subject must not be receiving chronic oral or intravenous steroids or immunosuppressive therapy.
14. Subjects must not be receiving medications that affect blood coagulation.
15. Subjects must not have had active cancer within the past year (other than adequately treated basal cell or squamous cell skin cancer) or require chemotherapy.
16. Subjects must not have uncontrolled insulin dependent diabetes mellitus.
17. Subjects who have had a seizure in the last two years will be excluded.
18. Subjects who have attempted suicide in the past 12 months will be excluded.
19. Subjects who are immunosuppressed or who have conditions that typically result in immunocompromise (including, but not limited to: ataxia-telangiectasia, cancer, Chediak-Higashi syndrome, combined immunodeficiency disease, complement deficiencies, DiGeorge syndrome, HIV/AIDS, hypogammaglobulinemia, Job syndrome, leukocyte adhesion defects, malnutrition, panhypogammaglobulinemia, Bruton disease, congenital agammaglobulinemia, selective deficiency of IgA and Wiscott-Aldrich syndrome) will be excluded.
20. Subjects with active psychiatric concerns, including but not limited to major depression, bipolar disorder, schizophrenia or other psychotic disorder and post-traumatic stress disorder. Individuals undergoing effective treatment for any of these disorders will not be excluded, but will be evaluated by a rehabilitation psychologist.
21. Subjects who report use of controlled, non-prescribed substances other than cannabis/marijuana will be excluded. If a subject reports use of cannabis, we will use the DAST-10 questionnaire to screen for level of abuse. An individual may be included if the score is 5 or less and if the neuropsychologist deems that they are eligible. Subjects reporting use of cannabis will also undergo a urine drug test to screen for other nonprescribed drugs. Subjects will be excluded if they test positive for any non-prescribed substance other than cannabis.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Explanted | 12 months
  Safety of the MIRA device will be measured by tracking the number of individuals explanted prior to the end of the study.

SECONDARY OUTCOMES:
Adverse Events | 12 months
  The type and frequency of device-related adverse events will be recorded by exams and check ins with participants during the study.
Peak-to-Peak Voltage | 12 months
  Peak-to-peak voltage will be measured over the study duration as a metric of signal quality.
Signal-to-Noise Ratio | 12 months
  Signal-to-noise ratio will be measured over the study duration as a metric of signal quality.
Device Control | 12 months
  Participants will be asked to make specific movements, which will be compared to target movements, in order to determine the ability to control different degrees of freedom. Performance will be measured over the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gaunt, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Ripple on a regular basis. All data will be de-identified. There is no definitive plan to share data with other researchers at this point in time.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Information will be shared throughout duration of collaboration with Ripple LLC.
Access Criteria: Collaborators will receive data and study materials according to existing data sharing agreements.